CLINICAL TRIAL: NCT04143308
Title: The Effects of Simultaneous Training of Walking and Cognitive Tasks on Cognitive Functions of People With Schizophrenia: the Development of Mobile Application System and Effectiveness Analysis
Brief Title: The Effects of Simultaneous Training of Walking and Cognitive Tasks on Cognitive Functions of People With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-SV(I)-20170080
Record Dates: First submitted 2019-10-18; First posted 2019-10-29 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia; Cognitive Function; Physical Activity; Quality of Life
Keywords: Schizophrenia; Cognitive functional training; Dual-task training; Aerobic exercise; Mobile application
MeSH Terms: conditions — Schizophrenia; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: We will conduct a single-blinded, randomized controlled study. Ninety participants will be randomly assigned to: simultaneous training of walking and cognitive group, the cognitive training group, and treatment as usual group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Simultaneous training of walking and cognitive group (Experimental): 1. Wearable technology (fitness wristband & App)
  2. SWATCH system (App & controller)
  3. 3 times a week (30 mins/ each time)
  4. Lasts for 12 weeks
  5. Simultaneous walking and cognitive training
  Interventions: Other: Simultaneous training of walking and cognitive group
- Cognitive training group (Active Comparator): 1. Wearable technology (fitness wristband & App)
  2. SWATCH system (App)
  3. 3 times a week (30 mins/ each time)
  4. Lasts for 12 weeks
  5. Cognitive training while sitting
  Interventions: Other: Cognitive training group
- Treatment as usual group (Active Comparator): 1. Keep treatment as usual group at health care system.
  Interventions: Other: Treatment as usual group

INTERVENTIONS:
Other: Simultaneous training of walking and cognitive group — Device:
  1. SWATCH system (App & controller)
  2. Wearable technology Fitness wristband & APP
  Arms: Simultaneous training of walking and cognitive group
Other: Cognitive training group — Device:
  1. SWATCH system (App)
  2. Wearable technology Fitness wristband & APP
  Arms: Cognitive training group
Other: Treatment as usual group — Keep treatment as usual
  Arms: Treatment as usual group

SUMMARY:
The object is to develop a training system of simultaneous walking and cognitive training for improving cognitive function of people with schizophrenia. The training program, called "Simultaneous Walk And Think for Cognitive Health mobile application software"(SWATCH App), is developed by researchers. A randomized controlled trial will be carried out to test the effectiveness of the training system. Ninety participants will be randomly assigned to: simultaneous training of walking and cognitive group, the cognitive training group, and treatment as usual group. The intervention for those groups will lasts for 12 weeks, with a 12 week of followup. The measurements include the cognitive function, physical fitness, and quality of life.

DETAILED DESCRIPTION:
Background: Schizophrenia is one of the severe mental disorders. In addition to psychiatric symptoms, cognitive impairment is a key clinical feature in this population, which significantly negatively influences their functional performance and independence. While the cognitive remediation therapy demonstrates positive results, it often involves specialized and expensive computerized cognitive training system, which limits its application in clinical setting. More evidence is available to support the benefits of exercise training on cognitive functions of schizophrenia. Combination of exercise and cognitive training is a promising program and can improve cognitive functions of the elderly. However, this combined therapy is still limited to schizophrenia. Simultaneous training of walking and cognitive tasks via auditory mobile application is an innovative program for saving cost, time, and manpower. Further study is needed to develop the simultaneous training program and to examine the effectiveness.

Purposes: To examine the effects of the training program on cognitive functions, fitness, functional performance and quality of life.

Methods: A 3-arm, single-blinded, randomized controlled trial is used to recruit 90 participants and then randomly allocated to the simultaneous training group, the cognitive training group, and the treatment as usual group. The first two training groups receive training for 30-40 minutes, 3 times a week for 12 weeks, as well as a follow-up of 12 weeks. All participants will be assessed at baseline, post-test and follow-up assessment. Primary outcome is cognitive function and secondary outcomes are fitness, functional performance, and quality of life.

Contribution: The study can be used as an evidence-based program to improve cognitive functioning of people with schizophrenia. With the development of mobile App and the use of fitness wearable device, the training program enables people with schizophrenia to walk and practice cognitive training simultaneously in a group format. It will help clinical professionals be able to serve the increasing number of people with severe mental illness with less manpower and specialized equipment. The study is also helpful to better understanding the isolated role of aerobic exercise in the dual-task training, and to apply to other groups, like the elderly or dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia or schizoaffective disorder by a psychiatric clinician on the basis of the criteria set the Diagnostic and Statistical Manual of Mental Disorders 5th edition, DSM-5, has been more than 1 year.
2. Age 20-60 years old.
3. Living in daycare center or community-based mental health rehabilitation services or rehabilitation ward.
4. Having stable psychiatric conditions (i.e., primary psychiatric medications had not changed for more than two months)
5. The MATRICS Consensus Cognitive Battery (MCCB) (Nuechterlein et al., 2008) shows that at least one domain with cognitive impairment (below the value of -1SD).
6. Can follow the research process and sign the consent form.

Exclusion Criteria:

1. Traumatic brain injury and other neurological diseases, alcohol and substance abuse
2. Pregnancy, cardiovascular disease, and unsuitable to exercise training due to physical movement difficulties
3. According participants' self-report, having following conditions, including severe heart failure, myocardial infarction, angina pectoris, chronic obstructive pulmonary disease, COPD, poor glycemic control (i.e., dialysis, diabetic neuropathy or retinopathy) and lower extremity arthritis
4. Uncontrolled hypertension with SBP> 160 mmHg or DBP> 110 mmHg
5. Diagnosis of intellectual disability
6. Unconscious or confusion of consciousness
7. Participating in other intervention studies

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  MATRICS Consensus Cognitive Battery: Traditional Chinese Version (MCCB) consists of 10 individually administered tests to measure cognitive performance in the following seven domains:
  1. Processing Speed
     1.1 Trail Making Test (TMT).
     1.2 Brief Assessment of Cognition in Schizophrenia: Symbol Coding (BACS SC).
     1.3 Category Fluency: Animal Naming (Fluency).
  2. Attention
     2.1 Continuous Performance Test: Identical Pairs (CPT-IP).
  3. Working memory
     3.1 Wechsler Memory Scale-III (WMS III): Spatial Span.
     3.2 Wechsler Letter: Number Sequencing (WAIS-III).
  4. Verbal Learning
     4.1 Hopkins Verbal Learning Test-Revised (HVLT-R).
  5. Visual Learning
     5.1 Brief Visuospatial Memory Test-Revised (BVMT-R).
  6. Reasoning and Problem Solving
     6.1 Neuropsychological Assessment Battery (NAB): Mazes.
  7. Social Cognition
  7.1 Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT): Managing Emotions.

SECONDARY OUTCOMES:
Body composition | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  Using Body Mass Index (BMI) as the measurement of body composition, which weight and height will be combined to report BMI in kg/m^2.
Cardiorespiratory fitness | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  Using 6-minute walk test (6MWT) as the measurement, which let the participant walks as far as possible over a total of six minutes on hard and flat floor. And the researcher will measure the distance that participant walks in 6 minutes.
Leg muscular strength and endurance | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  Using 30-Second Sit to Stand Test. The participant will sit in the middle of the chair, and rise to a full standing position, then sit back down again. Repeat these movements for 30 seconds. And researcher will count the times.
Balance and Agility | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  The Timed Up and Go test (TUG). It measures the time that the participant takes to rise from a chair, walk eight foots, turn around, walk back to the chair, and sit down.
Dual-Task Performance Involving Hand Dexterity and Cognitive Tasks | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  Dual-Task Performance Involving Hand Dexterity and Cognitive Tasks, this test is combine the Purdue Pegboard Test (PPT; Tifﬁn & Asher, 1948) and the Serial Sevens Subtraction Test (SSST; Manning, 1982), Purdue Pegboard Test use to measures hand dexterity; Serial Sevens Subtraction Test as a cognitive task for the dual-task condition.
Instrumental Activity of Daily Living (IADL) | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  Lawton and Brody Instrumental Activity of Daily Living Scale is a self-report survey. It is used to evaluate the degree of participant's instrumental activities. There are total 8 descriptions, the scale scores ranges is between 0 to 8. The higher values represent a better outcome.
Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) | Change from baseline outcome measure at 12th week (post-test), and at 24th week (follow-up test)
  Schizophrenia Quality of Life Scale Revision 4 is a self-report survey. It is used to evaluate the degree of participant's quality of life. There are total 33 items, the scale scores statements are rated 1 (never) to 5 (always). The higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-De Chen, Ph.D., Principal Investigator — Department of Occupational Therapy, College of Health Sciences, Kaohsiung Medical University
Locations (1):
- Ming-De Chen, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No